CLINICAL TRIAL: NCT06843239
Title: A Phase 2, Multi-Center Study Consisting of a Randomized, Double-Blind, Placebo-Controlled Period, Followed by an Open-Label Extension Period, to Assess the Efficacy, Safety, and Tolerability of Tibulizumab in Adults With Systemic Sclerosis
Brief Title: Tibulizumab Systemic Sclerosis Understanding and Response Evaluation (TibuSURE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zura Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZB-106-SS-201; 2024-519335-42-01 (EU CTIS Number)
Record Dates: First submitted 2025-02-07; First posted 2025-02-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Systemic Sclerosis (SSc); Scleroderma
Keywords: Scleroderma; Systemic Sclerosis (SSc); Tibulizumab; Cutaneous; Interstitial lung disease (ILD); Autoimmune diseases; Immune system diseases; Systemic Sclerosis interstitial lung disease (SSC-ILD); Skin Diseases
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Lung Diseases, Interstitial; Autoimmune Diseases; Immune System Diseases; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tibulizumab (Experimental): Subcutaneous injection
  Interventions: Biological: Tibulizumab
- Placebo (Placebo Comparator): Subcutaneous injection
  Interventions: Biological: Tibulizumab; Other: Placebo

INTERVENTIONS:
Biological: Tibulizumab — Anti BAFF/IL-17 antibody
  Other Names: ZB-106
Other: Placebo — Placebo (inactive)
  Other Names: ZB-106 placebo
  Arms: Placebo

SUMMARY:
The study is a Phase 2, multi-center, randomized, double-blind, placebo-controlled study to evaluate the effects of tibulizumab over 24 weeks (Period 1) in adult participants with systemic sclerosis, followed by an open-label extension period where all active participants will receive tibulizumab and will be evaluated for an additional 28 weeks (Period 2)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age
* Body mass index between 18.0 and 38.0 kg/m²
* Fulfills classification criteria for SSc according to ACR/EULAR 2013 criteria
* Has diffuse cutaneous SSc, defined as mRSS >0 over at least one skin area proximal to the elbows and/or knees, in addition to acral fibrosis
* Has had SSc (defined as the first non-Raynaud's phenomenon (RP) symptom or sign attributed to SSc) for ≤7 years
* mRSS ≥15 and ≤45 at screening. Additional requirements for participants ≥2 years to ≤7 years from SSc onset and RNA Polymerase III antibody positive
* FVC >50% predicted
* Diffusing capacity of the lungs for carbon monoxide (DLCO) ≥40% predicted (corrected for hemoglobin)

Exclusion Criteria:

* Has any of the following complications:

  * Left ventricular failure
  * Pulmonary arterial hypertension
  * Renal crisis within previous 6 months
  * Gastrointestinal dysmotility within previous 3 months
  * Digital ischemia with gangrene, amputation, or unscheduled hospitalization within previous 3 months
* Current rheumatic disease other than SSc that could interfere with assessment of SSc
* Lung disease requiring continuous oxygen therapy
* Evidence or suspicion of active or latent tuberculosis
* Active Crohn's Disease or ulcerative colitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
[Period 1] Change from baseline in modified Rodnan Skin Score (mRSS) at 24 weeks | Week 24
  The mRSS assesses skin thickness at 17 different cutaneous sites across the body using a scale from 0 (normal skin) to 3 (severe thickening), with a total score ranging from 0 (no thickening) to 51 (severe thickening in all 17 areas)
[Period 2] Safety and tolerability of tibulizumab | Week 52
  Assessed by the incidence of all treatment-emergent adverse events (TEAEs), as well as changes from baseline in vital signs, electrocardiogram (ECG) parameters, and laboratory results

SECONDARY OUTCOMES:
[Period 1] Change from baseline in quantitative interstitial lung disease (QILD) obtained with high-resolution quantitative tomography (HRCT) in the whole lung in participants with SSc-interstitial lung disease (ILD) | Week 24
  HRCT measures the extent of interstitial lung disease by quantifying the amount of lung fibrosis, ground-glass opacity, and honeycomb lung, which are used to calculate the QILD score (scores can range from 0 to 100%, with higher scores indicating greater disease extent)
[Period 1] Change from baseline in forced vital capacity (FVC) in participants with SSc-ILD | Week 24
  FVC is the amount of air that can be forcibly exhaled after the deepest possible breath
[Period 1] Change from baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) | Week 24
  HAQ-DI evaluates patients' self-assessed degree of disability across eight categories, with scores ranging from 0 to 3, where 3 indicates the worst degree of disability
[Period 1] Safety and tolerability of tibulizumab | Week 24
  Assessed by the incidence of all TEAEs, as well as changes from baseline in vital signs, ECG parameters, and laboratory results
[Period 2] Change from baseline in mRSS | Week 52
  The mRSS assesses skin thickness at 17 different cutaneous sites across the body using a scale from 0 (normal skin) to 3 (severe thickening), with a total score ranging from 0 (no thickening) to 51 (severe thickening in all 17 areas)
[Period 2] Change from baseline in QILD obtained with HRCT in the whole lung in participants with SSc-ILD | Week 52
  HRCT measures the extent of interstitial lung disease by quantifying the amount of lung fibrosis, ground-glass opacity, and honeycomb lung, which are used to calculate the QILD score (scores can range from 0 to 100%, with higher scores indicating greater disease extent)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Zura Bio Inc
Locations (51):
- United States (6):
  - UCSD Altman Clinical and Translational Research Institute Center for Clinical Research, La Jolla, California
  - IRIS Research and Development LLC, Plantation, Florida
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Rheumatology Associates, Arlington, Texas
- Argentina (11):
  - STAT Research S.A., Buenos Aires, Buenos Aires
  - Centro de Investigaciones Médicas Tucumán, San Miguel de Tucumán, Tucumán Province
  - Organización Médica de Investigación, Buenos Aires
  - Centro de Investigación y Prevención Cardiovascular-Arenales, Buenos Aires
  - Hospital General de Agudos Dr. José María Ramos Mejia, Buenos Aires
  - Instituto de Investigación Clínica TyT, Buenos Aires
  - Centro Medico de Estudios Clinicos y Farmacovigilancia (CECYF), Buenos Aires
  - Consultorios Médicos Dr. Doreski, Buenos Aires
  - Consultora Integral de Salud Centro Médico Privado, Córdoba
  - Instituto CER S.A., Quilmes
  - AES - AS - Clinica Mayo de Urgencias, San Miguel de Tucumán
- Chile (6):
  - CTR Estudios Clinicos, Santiago
  - Enroll SpA, Santiago
  - Centro de especialidades médicas Vanguardia, Temuco
  - Clinical Research Chile SpA, Valdivia
  - Centro de Estudios Clinicos Victoria Limitada (Cevic), Victoria
  - Dermacross Clinica Dermatologica, Vitacura
- Pécsi Tudomanyegyetem - Vasvari Pal u., Pécs, Hungary
- Mexico (5):
  - Mediadvance Clinical, Chihuahua City
  - PanAmerican Clinical Research, Guadalajara
  - Medical Care and Research S.A. de C.V., Mérida
  - Centro de Investigación y Tratamiento Reumatológico S.C, Miguel Hidalgo
  - Oaxaca Site Management Organization - Clinic - OSMO - PPDS, Oaxaca City
- Poland (7):
  - M2M Med-ul., Chorzów
  - Malopolskie Badania Kliniczne Sp. z o.o., Krakow
  - Malopolskie Centrum Kliniczne, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Twoja Przychodnia PCM - ul., Poznan
  - Klinika Reuma Park sp . zoo Sp.k., Warsaw
  - MICS Centrum Medyczne Warszawa, Warsaw
- Romania (3):
  - Center for Clinical and Basic Research (CCBR), Bucharest
  - Sf.Maria Clinical Hospital, Bucharest
  - Hiperdia Romania, Bucharest
- Serbia (2):
  - Institute of Rheumatology - PPDS, Belgrade
  - Military Medical Academy, Belgrade
- Spain (3):
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Corporacio Sanitaria Parc Tauli, Barcelona
  - Hospital Quironsalud Infanta Luisa, Seville
- United Kingdom (7):
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal National Hospital for Rheumatic Diseases, Bath
  - Ninewells Hospital, Dundee
  - Chapel Allerton Hospital, Leeds
  - Aintree University Hospital, Liverpool
  - Royal Free Hospital, London
  - Haywood Community Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://tibusure.patientwing.com/?campaignId=1796